CLINICAL TRIAL: NCT04759534
Title: Phase III Clinical Study to Evaluate the Efficacy and Safety of PCSK9 Inhibitors in the Prevention of Chinese Heterozygous Familial Hypercholesterolemia
Brief Title: Application of PCSK9 Inhibitors in Patients With Heterozygous Familial Hypercholesterolemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenzhen People's Hospital (Other)
Collaborators: Innovent Biopharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LQY-PCSK9-heterozygous
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Efficacy and Safety; Heterozygous Familial Hypercholesterolemia; PCSK9
Keywords: PCSK9 inhibitor; heterozygous familial hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Central laboratory uses random number table to generate random sequence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group 1 (Experimental): Received abdominal subcutaneous injection of IBI306 150 mg Q2W
  Interventions: Biological: protein convertase subtilisin/kexin type 9 inhibitor
- Treatment group 2 (Experimental): Received abdominal subcutaneous injection of IBI306 150 mg Q4W
  Interventions: Biological: protein convertase subtilisin/kexin type 9 inhibitor
- Placebo Group 1 (Placebo Comparator): Received a subcutaneous injection of placebo Q2W in the abdomen
  Interventions: Biological: protein convertase subtilisin/kexin type 9 inhibitor
- Placebo Group 2 (Placebo Comparator): Received a subcutaneous injection of placebo Q4W in the abdomen
  Interventions: Biological: protein convertase subtilisin/kexin type 9 inhibitor

INTERVENTIONS:
Biological: protein convertase subtilisin/kexin type 9 inhibitor — IBI306 is a kind of protein convertase subtilisin/kexin type 9 inhibitor.Received abdominal subcutaneous injection of IBI306 150 mg Q2W or 300 mg Q4W

SUMMARY:
This study plans to enroll several patients with heterozygous familial hypercholesterolemia, randomly assigned to different dose groups, and randomly receiving subcutaneous injection of IBI306150 mg or placebo every two weeks: or subcutaneous injection of IBI306 450mg every four weeks (n=49) or placebo (n=25) treatment, treatment lasted for 12 weeks. During randomization, the LDL-C level (<4.8mmol/L or ≥4.8mmol/L) observed during the screening period visit (VI), and whether ezetimibe was used for stratification. After 12 weeks, each group entered the 12-week open-period treatment, in which subjects in the IBI306 group continued to receive IBI306 treatment, and subjects in the placebo group stopped using placebo and received IBI306 treatment. The exploratory endpoint is the population pharmacokinetic characteristics of IBI306 in Chinese heterozygous familial hypercholesterolemia population.

DETAILED DESCRIPTION:
This study plans to enroll 148 patients with heterozygous familial hypercholesterolemia, and maintain a low-fat diet and stably take the current anterior-lowering therapy for at least 4 weeks. Randomly enter different dose groups at 1:1. 2: 1 randomized to receive subcutaneous injection of IBI306150 mg (n=49) or placebo (n=25) every two weeks: or subcutaneous injection of IBI306 450mg (n=49) or placebo (n=25) every four weeks , The treatment lasted 12 weeks. During randomization, the LDL-C level (<4.8mmol/L or ≥4.8mmol/L) observed during the screening period visit (VI), and whether ezetimibe was used for stratification. After 12 weeks, each group entered the 12-week open-period treatment, in which subjects in the IBI306 group continued to receive IBI306 treatment, and subjects in the placebo group stopped using placebo and received IBI306 treatment. The primary endpoint was the percentage change in LDL-C levels from baseline at 12 weeks. The secondary endpoints were the changes in blood lipid levels from baseline at 12 and 24 weeks, drug safety, and immunogenicity. The exploratory endpoint is the population pharmacokinetic characteristics of IBI306 in Chinese heterozygous familial hypercholesterolemia population. If necessary, the dose of IBI306 will be adjusted according to the results of the ongoing multi-dose climbing study. After the open period, the subjects will undergo an 8-week safety visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated informed consent form.
2. Men or women aged ≥18 and ≤80 at the time of screening.
3. Body weight ≥ 40 kg at the time of screening.
4. According to British Simon Broome (SBR) standards, HeFH is diagnosed or suspected:

   Diagnosis of HeFH: Total cholesterol> 7.5 mmol/L, or LDL-C concentration> 4.9 mmol/L, and at least one of the following two can be diagnosed: 1) The patient has tendon xanthoma, or his relatives (first-degree or At least one person at Level 2) has tendon xanthoma; 2) has evidence of LDL receptor, ApoB-100 or PCSK9 gene mutation; Suspected HeFH: Total cholesterol> 7.5 mmol/L, or LDL-C concentration> 4.9 mmol/L, and at least one of the following two is suspected HeFH: 1) Second-degree relatives before 50 years old or first-degree relatives 60 years old Previous history of myocardial infarction; 2) First-degree or second-degree adult relatives have a history of total cholesterol>7.5mmol/L or children, brothers, sisters have a history of total cholesterol>6.7mmol/L before the age of 16 or 16 years old.
5. Maintain a low-fat diet and stably take the current lipid-lowering therapy (taking moderate-intensity or above statins, except for statin intolerance, with or without ezetimibe, niacin, and omega fatty acids) for at least 4 weeks. If you are taking fibrates, the fibrates are treated stably for at least 6 weeks.
6. The fasting LDL cholesterol concentration of patients with a history of atherosclerotic cardiovascular disease at the time of screening was ≥1.8 mmol/L; the fasting LDL cholesterol concentration of patients without a history of atherosclerotic cardiovascular disease was ≥2.6 mmol/L.
7. The subject indicated that they are willing and cooperate to complete all the steps in the study and the study intervention period.

Exclusion Criteria:

1. Patients diagnosed as homozygous familial hypercholesterolemia.
2. He had undergone dialysis or plasma exchange within 4 months before screening.
3. Patients who have received liver transplant surgery in the past.
4. Adjust the treatment plan or dose of statins, ezetimibe, niacin, and omega fatty acids within 4 weeks before the screening of subjects (these subjects can stabilize the current lipid-lowering drug dosage for 1 month, and then Re-filter).
5. New York Heart Association (NYHA) grade III or IV heart failure, or recently detected left ventricular ejection fraction ≤ 30%.
6. Poorly controlled severe arrhythmia, defined as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation with rapid ventricular rate or supraventricular tachycardia.
7. Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass grafting or stroke occurred within 3 months before enrollment.
8. Plan to perform percutaneous coronary intervention, coronary artery bypass grafting or other heart surgery during the study period.
9. Type 1 diabetes or poor blood sugar control (HbA1c>8.5%), or type 2 diabetes requiring multiple injections of insulin daily.
10. There are uncontrolled clinical diseases that may affect blood lipids or lipoprotein levels (in patients with thyroid hormone replacement therapy, the thyroid hormone dose needs to be stable for at least 6 weeks before the screening visit). Poorly controlled hypothyroidism or hyperthyroidism is defined as TSH <the lower limit of normal, or> 1.5 times the upper limit of normal.
11. Poorly controlled hypertension is defined as a sitting systolic blood pressure> 180 mmHg or diastolic blood pressure> 110 mmHg confirmed by repeated measurements.
12. Moderate to severe renal insufficiency, defined as the estimated glomerular filtration rate <30 ml / min / 1.73 m2 during the screening period.
13. Active liver disease or liver function impairment is defined as the screening period determined by local laboratory analysis, aspartate aminotransferase or alanine aminotransferase> 3 times the upper limit of normal (ULN).
14. Creatine kinase (CK) ≥ 3 times of ULN during screening.
15. As judged by the investigator, there is a known active infection or major blood, kidney, metabolic, gastrointestinal, or endocrine dysfunction.
16. Once diagnosed with deep vein thrombosis or pulmonary embolism.
17. Except for those who have been sterilized or menopausal, female subjects with potential for pregnancy, if they are unwilling to inform their sexual partners that they will participate in the clinical study, and take effective measures during the use of the study drug and within 15 weeks after the last dose of the study drug Contraceptive measures. Male subjects are unwilling to inform their female sexual partners that they participate in the clinical study.
18. Subjects who are pregnant or breastfeeding, or plan to become pregnant or breastfeeding during the period of study medication or within 15 weeks after the last dose of study medication.
19. Suffered from malignant tumors in the past 5 years (except for non-melanoma skin cancer, cervical carcinoma in situ, ductal carcinoma in situ of the breast or stage 1 prostate cancer).
20. The subject has received PCSK9 inhibitor treatment or participated in other studies that inhibit PCSK9.
21. Known allergy to study drug and its ingredients.
22. Those who are judged by the investigator to be unsuitable to participate in the study (for example, alcohol or other drug abuse, inability or unwillingness to comply with the agreement, or mental illness).
23. Currently participating in another medical device or drug research, or the previous medical device or drug clinical research has ended, or receiving other research drugs for less than 30 days.
24. In any other circumstances, the investigator or sponsor believes that it may impair the subject's ability or safety to give written informed consent and/or comply with all necessary research procedures.
25. Human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibodies, HIV or syphilis antibodies were positive at the time of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
LDL-C | 12 weeks after baseline
  Percentage decrease in LDL-C from baseline
LDL-C | 24 weeks after baseline
  Percentage decrease in LDL-C from baseline
non HDL-C | 12 weeks after baseline
  Percentage decrease in non HDL-C from baseline
non HDL-C | 24 weeks after baseline
  Percentage decrease in non HDL-C from baseline
ApoB | 12 weeks after baseline
  Percentage decrease in ApoB from baseline
ApoB | 24 weeks after baseline
  Percentage decrease in ApoB from baseline

SECONDARY OUTCOMES:
safty | 12 weeks after baseline
  From the first administration to the last visit, the incidence of adverse events;
safty | 24 weeks after baseline
  From the first administration to the last visit, the incidence of adverse events;

CONTACTS AND LOCATIONS:
Overall Officials: dong shaohong, doctor, Study Chair — Shenzhen People's Hospital
Locations (1):
- xili People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No